CLINICAL TRIAL: NCT00054548
Title: A Phase I Study of Antisense Bcl-2 Oligonucleotide (G3139) in Combination With Carboplatin and Paclitaxel in Patients With Advanced Solid Tumors
Brief Title: Combination Chemotherapy Plus Oblimersen in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00010; CO 02904; NCI-5912; WCCC-CO-02904; U01CA062491 (NIH)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — oblimersen; Paclitaxel; Taxes

ARMS (1):
- Treatment (oblimersen sodium, paclitaxel) (Experimental): Patients receive oblimersen IV continuously on days 1-7 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of oblimersen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  An additional cohort of 12-15 patients receives treatment as above with oblimersen at the MTD.
  Interventions: Biological: oblimersen sodium; Drug: paclitaxel; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase I trial to study the effectiveness of combining carboplatin and paclitaxel with oblimersen in treating patients who have advanced solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Oblimersen may increase the effectiveness of carboplatin and paclitaxel by making tumor cells more sensitive to the drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of G3139 in combination with carboplatin and paclitaxel.

II. To determine the quantitative and qualitative nature of toxicities of G3139 with carboplatin and paclitaxel.

III. To measure G3139 activity in peripheral blood lymphocytes by quantitating Bcl-2/Bax expression and transcription, as well as T-cell functioning and signaling.

IV. To measure G3139 activity in tumor biopsy specimens by quantitating Bcl-2/Bax expression and transcription.

V. To determine the pharmacokinetics of carboplatin, paclitaxel, and G3139, as well as intratumoral G3139 levels.

VI. To screen various signal transduction pathways that may be affected by Bcl-2 down-regulation in PBMC and tumor biopsy specimens in order to better understand the mechanism of G3139 chemosensitization.

VII. To seek preliminary evidence of antitumor activity for the combination of G3139, carboplatin, and paclitaxel.

OUTLINE: This is a dose-escalation study of oblimersen.

Patients receive oblimersen IV continuously on days 1-7 and paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of oblimersen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

An additional cohort of 12-15 patients receives treatment as above with oblimersen at the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed solid malignancy that is metastatic or unresectable and for which no standard curative therapy exists; patients with lymphoma are excluded
* ECOG performance status 0, 1, or 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for three months after discontinuation of treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients will need to have a central line or nurse-placed PICC line in place prior to treatment on the protocol

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases will be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to G3139 or other agents used in study, unless approved by investigator
* No pre-existing grade >= 2 neuropathy
* No personal history of a bleeding diathesis given potential significant antiplatelet effects of therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with G3139
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2002-10; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) defined as the highest safely tolerated dose where at most 1 patient experiences a dose-limiting toxicities (DLT) and the next higher dose having at least 2 patients who experience DLT | 21 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters of G3139 in combination with paclitaxel and carboplatin | Day 1, 4, 5, and 6 of course 1
  All PK parameters will be summarized by dose level with simple summary statistics: means, medians, ranges, and standard deviations (if numbers and distribution permit).
Disease response as having either progressive disease (PD), stable disease (SD), a partial response (PR), or a complete response (CR) | Up to 6 years
  Disease response will be summarized in tabular format showing the number and percent of patients in each category/dose level. Dose-response relationships will be explored by logistic regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States